CLINICAL TRIAL: NCT01919710
Title: Phase 1 Study of rHSA/GCSF in Neutropenia After Chemotherapy of Cancer Patients
Brief Title: Safety and Efficacy Studies of rHSA/GCSF Fusion Protein For Injection to Treat Neutropenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin SinoBiotech Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9314-rHSA/GCSF; 2011L01837 (Registry Identifier: China SFDA#2011L01837)
Record Dates: First submitted 2012-11-26; First posted 2013-08-09 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Underdose (Unintentional); Cancer; Tumor
Keywords: Neutropenia; chemotherapy; rHSA/GCSF
MeSH Terms: conditions — Neoplasms; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rHSA/GCSF for injection (Experimental): rHSA/GCSF Start from 300mcg
  Interventions: Drug: rHSA/GCSF

INTERVENTIONS:
Drug: rHSA/GCSF — for treatment of neutropenia
  Other Names: Long acting rhG-CSF fusion protein

SUMMARY:
Safety and efficacy studies of rHSA/GCSF fusion protein for injection in treatment of neutropenia induced by chemotherapy of cancer patients.

DETAILED DESCRIPTION:
A dosage climbing for the safety and efficacy studies for the neutropenia induced by chemotherapy cancer patients Repeat-dose studies for the safety and efficacy studied for the neutropenia.

ELIGIBILITY:
Inclusion Criteria:

- chemotherapy induced neutropenia

Exclusion Criteria:

- treated with other biological drugs or other neutropenia therapy drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 14 days
  Number of participants with adverse events as a measure for safety and tolerability after single and multiple dose of rHSA/GCSF

SECONDARY OUTCOMES:
AUC | 14 days
  AUC after single and multiple dose of rHSA/GCSF

CONTACTS AND LOCATIONS:
Overall Officials: Jun ZHU, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China